CLINICAL TRIAL: NCT06035172
Title: The Effect of Guided Imagery and Music Play on Labor Pain, Anxiety, and Birth Experience: A Randomized Controlled Study
Brief Title: The Effect of Guided Imagery and Music Play on Labor Pain, Anxiety, and Birth Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/362
Record Dates: First submitted 2023-07-11; First posted 2023-09-13 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-05

CONDITIONS: Labor Pain
Keywords: Birth pain; music listening; positive birth; guided imagery
MeSH Terms: conditions — Labor Pain | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- guided imagery group (Experimental)
  Interventions: Behavioral: guided imagery
- music group (Experimental)
  Interventions: Behavioral: music recital
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: guided imagery — The guided imagery technique, which is one of these methods, is used in the method of pain by establishing a connection between mind and body. In the technique, a peaceful scene is depicted in which positive energy is reflected in the person to ensure complete relaxation and relaxation.
  Arms: guided imagery group
Behavioral: music recital — It is stated that the acemasiran tune (instrumental music) has a reducing effect on the duration of labor, as well as having labor pain and muscle relaxant properties.
  Arms: music group

SUMMARY:
Purpose: The aim of this project is to examine the effects of guided imagery and music performance during labor on labor pain, anxiety and birth experience.

Methods: The research to be carried out within the scope of the project is randomized controlled and has an experimental research design. The population of the research consists of primiparous pregnant women who applied to the Istanbul Provincial Health Directorate, Istanbul Training and Research Hospital, Suleymaniye Obstetrics and Pediatrics Additional Service Building, Birth Unit. Eligible participants in the study sample will be randomly selected at a 1:1:1 ratio. In the calculation of the sample size, using the G*Power (3.1.9.2) program, 5% first type error, 0.30 standardized effect size, distribution ratio to 1 groups, 90% power considering data loss, and the minimum sample size required for 3 groups was 144 people in total. calculated as 48 cases for each group. The group of pregnant women who meet the inclusion criteria will be determined by using the "Randomizer.org" program. In this direction, 48 people (guided imagery) should be included in experiment 1, 48 people in experiment 2 (musical concert) and 48 people in control group. "Informed Consent Form" and "Voluntary Consent Form" will be presented to the pregnant women included in the study, by giving information about the study."Personal Information Form", "Visual Analogue Scale (VAS)", "State Trait Anxiety Scale (STAI Form TX-1)" and "Birth Expectations and Experiences Scale-Part 1 (DBSS-1)" will be applied to pregnant women assigned to the Guided Imagery Group. . In the active phase of labor, when the cervical opening is measured as 4-5 cm, 6-7 cm and 8-10 cm, a 15-minute guided imagery concert (of the scenario determined for the birth process) prepared by the researchers within the scope of the literature, with the service of a ney artist and a psychological counselor, is played by bluetooth from an MP3 player. The pregnant woman will be listened to by the researcher through headphones. "VAS" will be applied after each attempt. 1 hour after the birth of the baby and placenta, data will be collected by applying "VAS", "STAI Form TX-1" and "Birth Expectations and Experiences Scale-Part 2 (DBSS-2)".

"Personal Information Form", "VAS", "STAI Form TX-1" and "DBSS-1" will be applied to pregnant women assigned to the music concert group. In the active phase of labor, when the cervical opening is measured as 4-5 cm, 6-7 cm and 8-10 cm, the 15-minute ney concert in the acemasiran tune (instrumental music), which was prepared by the researchers with the service of the ney artist within the scope of the literature (the scenario determined for the birth process), was played from the MP3 player via bluetooth headphones. The pregnant woman will be listened to by the researcher. "VAS" will be applied after each attempt. Data will be collected by applying "VAS", "STAI Form TX-1" and "DBSS-2" 1 hour after the birth of the baby and placenta.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35,
* Primiparous and singleton pregnancy,
* No risky pregnancy,
* At 38 to 42 weeks of pregnancy,
* Being literate and able to speak and understand Turkish,
* Pregnant women with a cervical dilation of 4 to 5 cm.

Exclusion Criteria:

* Being under the age of 18,
* Presence of chronic disease,
* Women who became pregnant as a result of the application of assisted reproductive techniques,
* Hearing problem,
* Having a known diagnosis of serious psychiatric illness.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Reduction of labor pain | 15 minutes
  labor pain assessed by VAS
Reduction of Anxiety | 15 minutes
  anxieties of vaginal birth assessed by STAI Form TX-1

CONTACTS AND LOCATIONS:
Locations (1):
- Betül Uncu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biana CB, Cecagno D, Porto AR, Cecagno S, Marques VA, Soares MC. Non-pharmacological therapies applied in pregnancy and labor: an integrative review. Rev Esc Enferm USP. 2021 Apr 16;55:e03681. doi: 10.1590/S1980-220X2019019703681. eCollection 2021. English, Portuguese. PMID 33886910
- [Background] Rantala A, Hakala M, Polkki T. Women's perceptions of the pain assessment and non-pharmacological pain relief methods used during labor: A cross-sectional survey. Eur J Midwifery. 2022 Apr 13;6:21. doi: 10.18332/ejm/146136. eCollection 2022. PMID 35515089
- [Background] Smith CA, Levett KM, Collins CT, Armour M, Dahlen HG, Suganuma M. Relaxation techniques for pain management in labour. Cochrane Database Syst Rev. 2018 Mar 28;3(3):CD009514. doi: 10.1002/14651858.CD009514.pub2. PMID 29589650
- [Background] Mirghafourvand M, Mohammad Alizadeh Charandabi S, Ghanbari-Homayi S, Jahangiry L, Nahaee J, Hadian T. Effect of birth plans on childbirth experience: A systematic review. Int J Nurs Pract. 2019 Aug;25(4):e12722. doi: 10.1111/ijn.12722. Epub 2019 Jan 24. PMID 30675962
- [Background] Kacar N, Ozcan Keser N. Comparison of the effect of mechanical massage and warm mechanical massage application on perceived labor pain and childbirth experience: A randomized clinical trial. Eur J Midwifery. 2021 Feb 27;5:5. doi: 10.18332/ejm/132883. eCollection 2021. PMID 33655203